CLINICAL TRIAL: NCT01482871
Title: Safety Study of ALG 1001 to Treat Diabetic Macular Edema
Brief Title: Safety Study of ALG- 1001 to Treat Diabetic Macular Edema
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allegro Ophthalmics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Focus 2
Record Dates: First submitted 2011-11-28; First posted 2011-12-01 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema
MeSH Terms: interventions — risuteganib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1.5 mg ALG-1001 (Experimental): Group Using 1.5 mg per 100 ul of ALG-1001
  Interventions: Drug: ALG-1001
- Arm 2.5 mg ALG-1001 (Experimental): Group Using 2.5 mg per 100 ul of ALG-1001
  Interventions: Drug: ALG-1001
- Arm 5.0 mg ALG-1001 (Experimental): Group Using 5.0 mg per 100 ul of ALG-1001
  Interventions: Drug: ALG-1001
- Arm 7.5 mg ALG-1001 (Experimental): Group Using 7.5 mg per 100 ul of ALG-1001
  Interventions: Drug: ALG-1001

INTERVENTIONS:
Drug: ALG-1001 — 1.5 mg per 100ul injected in the eye on day 0, day 30 and day 60 and followed for 180 days until unacceptable toxicity develops
  Arms: Arm 1.5 mg ALG-1001
Drug: ALG-1001 — 2.5 mg per 100ul injected in the eye on day 0, day 30 and day 60 and followed for 180 days until unacceptable toxicity develops
  Arms: Arm 2.5 mg ALG-1001
Drug: ALG-1001 — 5.0 mg per 100ul injected in the eye on day 0, day 30 and day 60 and followed for 180 days until unacceptable toxicity develops
  Arms: Arm 5.0 mg ALG-1001
Drug: ALG-1001 — 7.5 mg per 100ul injected in the eye on day 0, day 30 and day 60 and followed for 180 days until unacceptable toxicity develops
  Arms: Arm 7.5 mg ALG-1001

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of ophthalmic intravitreal injection of ALG - 1001 in human subjects with diabetic macular edema. The primary endpoint of this study is observation of dose limiting toxicity and maximum tolerated dose. The secondary endpoint of this study is observation of a clinical effect in BCVA (ETDRS letters) and OCT central macular thickness.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety and efficacy of ophthalmic intravitreal injection of ALG - 1001 in human subjects with diabetic macular edema. The primary endpoint of this study is observation of dose limiting toxicity and maximum tolerated dose. The secondary endpoint of this study is observation of a clinical effect in best corrected visual acuity (BCVA) (ETDRS letters) and OCT central macular thickness.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18 years of age or older.
2. Patient (male or female) with active diabetic macular edema (DME).
3. Patient whose study eye has a best corrected visual acuity (BCVA) of 20/50 to 20/160 ETDRS equivalent (65 letters to 36 letters), that in the opinion of the investigator is primarily due to DME will be intravitreally injected with 0.10 cc containing 1.5mg/100µl or 2.5mg/100µl of ALG-1001. Decrease in BCVA must be assessed based on clinical exploration, macular thickening, presence of clinical significant macular edema and/or OCT findings consistent with diabetic macular edema.
4. Patient whose study eye has a best corrected visual acuity (BCVA) of 20/200 or worse ETDRS equivalent (35 letters or less), that in the opinion of the investigator is primarily due to DME will be intravitreally injected with 0.10 cc containing 5.0mg/100µl or 7.5mg/100µl of ALG-1001. Decrease in BCVA must be assessed based on clinical exploration, macular thickening, presence of clinical significant macular edema and/or OCT findings consistent with diabetic macular edema.
5. Patients Intra-Ocular Pressure (IOP) is under control, IOP ≤ 25 mm
6. Patient is willing and able to return for all study visits.
7. Patient is able to meet the extensive post-op evaluation regimen
8. Patient can understand and sign Informed Consent form.

Exclusion Criteria:

* 1. Patients with Media Opacities or abnormalities that would preclude observation of the Retina.

  2. Patients with active Proliferative Diabetic Retinopathy (PDR) in the study eye such as NVE, NVD, Vitreous Hemorrhage, or Neovascular Glaucoma.

  3. Patients with current or prior Retinal Detachments, Retinal tears, or Tractional Detachments in either eye.

  4. Patients with significant epiretinal membranes determined by the investigator to be contributing to the macular edema.

  5. Patients with other retinal pathologies that would interfere with their vision.

  6. Patient that has Chronic or Recurrent Uveitis. 7. Patient that has undergone Vitrectomy (anterior or pars plana) in the study eye.

  8. Patient has ongoing Ocular infection or inflammation in either eye. 9. Patient has a history of intravitreal injections of any type in the study eye within the last 45 days prior to study enrollment.

  10. Patient has a history of focal laser of any type in the study eye within the last 90 days prior to study enrollment.

  11. Patient has a history of cataract surgery complications/vitreous loss in the study eye.

  12. Patient has congenital eye malformations in the study eye. 13. Patient has a history of penetrating Ocular Trauma in the study eye. 14. Patient is mentally handicapped. 15. Patient is Pregnant or Nursing female. If subject is 18 to 60 years old. Negative pregnancy test during the screening window.

  16. Patient that is currently participating in any other Clinical Research Study 17. Patient has contraindication to the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Observation of dose limiting toxicity | 6 months
  The primary endpoint of this study is observation of dose limiting toxicity and the maximum tolerated dose. This determination will be made by the following criteria : Ocular Adverse Events by standard Clinical Ophthalmic examination Visual acuity changes from BCVA (ETDRS equivalent) at baseline by Slit Lamp Bio-microscopy, Tonometry, Indirect Ophthalmoscopy/ Fundus Photography, Fluorescein Angiography, OCT Central Macular Thickness, and ERG Examination

SECONDARY OUTCOMES:
Improvements in BCVA ETDRS | 6 months
  Reduction in OCT central macular thickness in subjects with baseline diabetic macular edema and Improvements in BCVA ETDRS letters at 4 meters from baseline to 30 days, 60 days and 90 days post injection evaluations with safety evaluations to 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Quiroz, M.D, Principal Investigator — Denver Medical Hospital
Locations (1):
- Apec Hospital La Ceguera, Mexico City, Mexico